CLINICAL TRIAL: NCT01942746
Title: Placebo-controlled Cross-over Studies Examining Blueberries Effects on Dark Vision and Recovery After Photo-bleaching
Brief Title: Blueberry Effects on Dark Vision and Glare Recovery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Atlantic Food and Horticulture Research Center (Other Government)
Collaborators: Dalhousie University (Other); U.S. Highbush Blueberry Council (Other)
Responsible Party: Principal Investigator, Wilhelmina Kalt, Scientist, Atlantic Food and Horticulture Research Center
Allocation: Non-Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: Blueberries and Vision
Record Dates: First submitted 2013-05-23; First posted 2013-09-16 (Estimated); Last update posted 2013-09-16 (Estimated); Status verified 2013-09

CONDITIONS: Blindness and Low Vision
Keywords: blueberry; anthocyanin; dark vision; photo bleaching; Visual Perception; Photic Stimulation
MeSH Terms: conditions — Blindness; Vision, Low | interventions — blueberry extract; Epinephrine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Blueberry Juice (Active Comparator): Commercially prepared single strength blueberry juice which was composed of a 50:50 blend of two highbush blueberry species (Vaccinium corymbosum L. 'Rubel' and V. ashei Reade 'TifBlue'). Volunteers consumed 300 mls of juice/day (247-271 mg anthocyanins (as C3G) daily) while on this intervention, for either 3 weeks (Blueberry Juice S2) or 12 weeks (Blueberry Juice L1).
  Interventions: Dietary Supplement: Blueberry Juice S2; Dietary Supplement: Blueberry Juice L1
- Blueberry Capsules (Active Comparator): Commercially prepared single strength blueberry juice which was composed of a 50:50 blend of two highbush blueberry species (Vaccinium corymbosum L. 'Rubel' and V. ashei Reade 'TifBlue')was freeze dried to a powder and encapsulated in gelatin capsules (Blueberry Capsules S2). Volunteers consumed 3 capsules/daily (7.11mg anthocyanin (as C3G eq) for 3 weeks.
  Interventions: Dietary Supplement: Blueberry Capsules S2
- Placebo (Placebo Comparator): Volunteers consumed in S2 three placebo capsules daily for 3 weeks. In L1 volunteers consumed 300ml placebo juice for twelve weeks. Placebo products contained no anthocyanins.
  Interventions: Dietary Supplement: Placebo Capsule S2; Dietary Supplement: Placebo Juice L1
- Washout (S2 and L1) (No Intervention): Washout periods involved no study products. Washout was 3 weeks in S2 and or 8 weeks (L1) in duration.

INTERVENTIONS:
Dietary Supplement: Blueberry Juice S2 — Blueberry Juice S2 was commercially prepared single strength blueberry juice composed of a 50:50 blend of Rubel (Vaccinium corymbosum L.) and Tifblue (Vaccinium ashei Reade) cultivars. Colorimetric analysis showed that S2 juice contained 6.04 (SD=0.20) mg anthocyanins (C3G) eq/g dry mass.
  Other Names: Single-strength blueberry juice, commercially prepared
  Arms: Blueberry Juice
Dietary Supplement: Blueberry Capsules S2 — Commercially prepared single strength blueberry juice composed of a 50:50 blend of Rubel (Vaccinium corymbosum L.) and Tifblue (Vaccinium ashei Reade) cultivars was freeze dried then powdered and encapsulated in gelatin capsules. Colorimetric analysis indicated an anthocyanin concentration in the powder of 2.37(SD=0.18) mg C3G eq per capsule.
  Other Names: freeze-dried blueberry juice powder
  Arms: Blueberry Capsules
Dietary Supplement: Placebo Capsule S2 — Placebo Capsule S2 (containing no anthocyanins) were prepared by freeze drying red beets and grinding them to fine powder before encapsulating in gelatine capsules. Red beets do not contain anthocyanins.
  Other Names: Red beet powder
  Arms: Placebo
Dietary Supplement: Placebo Juice L1 — Placebo juice was prepared from water, sugars, citric acid, sodium citrate, and artificial colors and flavours, then pasteurized. The placebo juice contains no anthocyanins.
  Arms: Placebo
Dietary Supplement: Blueberry Juice L1 — Blueberry Juice L1 was commercially prepared single strength blueberry juice composed of a 50:50 blend of Rubel (Vaccinium corymbosum L.) and Tifblue (Vaccinium ashei Reade) cultivars. Colorimetric analysis showed that L1 juice contained 6.83 (SD=0.20) mg cyanidin-3-glucoside equivalents (C3GE)/g dry mass at the start of the study, declining to 5.52 (SD=0.09) mg C3GE/g dry mass after 3 months refrigerated storage.
  Other Names: single strength blueberry juice, commercially prepared
  Arms: Blueberry Juice

SUMMARY:
Clinical evidence for effects of plant anthocyanins on vision, and particularly night vision is controversial. Two clinical trials were conducted to investigate whether blueberry juice consumption affected visual dark adaptation, functional night vision, and recovery after photo-bleaching of the retina. One trial (S2) employed a 3 week intervention and washout period, and two doses of blueberries plus a placebo. The other trial (L1) employed a 12 week intervention plus an 8 week washout and tested one blueberry juice dose against a juice placebo.

DETAILED DESCRIPTION:
Vision Tests: 1. Dark adaptometry, 2. scotopic visual acuity, 3. scotopic contrast sensitivity, 4. rod/cone conversion, 5. recovery after retinal photobleaching

ELIGIBILITY:
Inclusion Criteria:

* visual acuity better than 6/7.5 on EDTRS acuity chart at 2.5m
* visual contrast sensitivity within normal range at 2.5m as tested on Visteck 3000
* stereo acuity better than 80 seconds of arc on Frisby stereoacuity test
* no ocular history other than refractive glasses
* no family history of eye disease

Exclusion Criteria:

* family history of retinal degeneration, glaucoma, diabetes, hypertension, cataract, or amblyopia (dimness in vision).
* evidence in subject (upon examination) of amblyopia (dimness in vision), manifest strabismus (unable to focus both eyes on one spot), or anisotropia (non-uniform responsiveness between both eyes).
* intraocular pressure above 21mmHG from an average of three measures using Mentor tonopen-XL

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2005-07; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Rate of vision adaptation to low light after blueberry juice and placebo ingestion for 3 weeks (S2). | Pre-intervention, and changes after 3 weeks of intervention, and again after 3 weeks of washout
  Effect of blueberry products and placebo on the rate of vision adaptation to low light. The rate of vision adaptation is measured by lowest perceptible light intensity after 30 min of darkness (dark threshold); time to reach dark threshold (min); time to reach rod/cone transition (min) [Time Frame: Pre-intervention, after 3 weeks intervention, again after a 3 week washout.] [Designated as safety issue: No]
Rate of vision adaptation to low light after ingestion of blueberry juice and placebo for 12 weeks (L1). | Preintervention, and changes after 8 and 12 weeks of intervention and after 4 and 8 weeks of washout
  Effect of blueberry products and placebo on the rate of vision adaptation to low light. The rate of vision adaptation is measured by lowest perceptible light intensity after 30 min of darkness (dark threshold); time to reach dark threshold (min); time to reach rod/cone transition (min) [Time Frame: Pre-intervention, after 8 and 12 weeks intervention, and again after 4 and 8 weeks washout] [Designated as safety issue: No]

SECONDARY OUTCOMES:
Rate of recovery of visual acuity after retinal photostress (S2). | Pre-intervention testing and testing for changes after 3 weeks of intervention and 3 weeks of washout
  After dark adaptation testing (primary outcome) and contrast sensitivity and visual acuity testing (other pre-specified outcome measures), participants are subjected to photostress of the retina using bright light. The time (sec) required to recover pre-stress acuity is measured.
Rate of recovery of visual acquity after retinal photostress (L1). | Pre-intervention and then testing for changes after 8 and 12 weeks of intervention and 4 and 8 weeks of washout.
  After dark adaptation testing (primary outcome) and contrast sensitivity and visual acuity testing (other pre-specified outcome measures) participants are subjected to photostress of the retina using bright light. The time (sec) required to recover pre-stress acuity is measured.

OTHER OUTCOMES:
Visual acuity and contrast sensitivity testing after dark adaptation (S2). | Testing preintervention and testing for changes after 3 weeks of intervention and 3 weeks of washout
  After dark adaptation testing (primary outcome measure) and before measuring rate of recovery from photo stress (secondary outcome) visual acuity in darkness and contrast sensitivity in darkness was measured using defined optotypes with different degrees of crowding and contrast. Performance was defined as the number of correct answers in 12 tests of acuity and 8 tests of contrast sensitivity.
Visual acuity and contrast sensitivity testing after dark adaptation (L1). | Testing preintervention and testing for changes after 8 & 12 weeks of intervention and 4 & 8 weeks of washout
  After dark adaptation testing (primary outcome measure) and before testing rate of recovery from photo stress (secondary outcome) visual acuity in darkness and contrast sensitivity in darkness was measured using defined optotypes with different degrees of crowding and contrast. Performance was defined as the number of correct answers in 12 tests of acuity and 8 tests of contrast sensitivity.

CONTACTS AND LOCATIONS:
Overall Officials: Wilhelmina Kalt, PhD, Principal Investigator — Agriculture and Agri-Food Canada; Francois Tremblay, PhD, Principal Investigator — Dalhousie University and IWK Health Center
Locations (1):
- Atlantic Food and Horicultural Research Center, Kentville, Nova Scotia, Canada

REFERENCES:
- [Derived] Kalt W, McDonald JE, Fillmore SA, Tremblay F. Blueberry effects on dark vision and recovery after photobleaching: placebo-controlled crossover studies. J Agric Food Chem. 2014 Nov 19;62(46):11180-9. doi: 10.1021/jf503689c. Epub 2014 Nov 6. PMID 25335781